CLINICAL TRIAL: NCT01926600
Title: Sublingual Administration is More Fast Than Oral or IV Administration in PPI Dosing With Respect to Intragastric pH and Therapeutic Effectiveness: a Prospective, Randomized, Controlled Trial
Brief Title: Sublingual Administration of PPI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jin Il Kim, MD, PhD, The Catholic University of Korea
Other Study IDs: 24 hour pH
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Gastric or Duodenal Ulcer
Keywords: gastric ulcer; duodenal ulcer; re-bleeding rate; intragastric pH; proton pump inhibitor
MeSH Terms: conditions — Duodenal Ulcer; Stomach Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PO: administrated by per oral
- IV: Administrated by intravenous
- SL: administrated by sublingual

SUMMARY:
Compare 24-hour intragastric pH and therapeutic effectiveness of proton pump inhibitor (PPI) among different administration methods: per oral (PO), intravenous (IV), and sublingual (SL).

DETAILED DESCRIPTION:
Intragastric pH and therapeutic effectiveness of PPI was compared among patients given PPI with different administration methods. 24 hour intragastric pH catheter was inserted in stomach of patients with peptic ulcer an hour prior to PPI administration in order to observe the initial change in pH. Three groups of patients were given PPI through per oral, intravenous, and sublingual administration methods. The hypothesis of this study is that sublingual administration will be faster than oral or IV administration in PPI dosing with respect to intragastric pH change and re-bleeding rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peptic ulcer disease
* Age: 20-75 years old
* Patients who submitted informed consent

Exclusion Criteria:

* Peptic ulcer disease with spurting and oozing
* Shock, hypotension, pregnancy
* Gastrointestinal malignancy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3 groups, each group with 20 subject with peptic ulcer ages between 20 to 75
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Measure 24-hour intragastric pH | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- St.Mary's Hopspital of the Catholic University, Seoul, South Korea